CLINICAL TRIAL: NCT03332394
Title: Impact of Goal-Directed COPD Care Model on Clinical and Patient-Reported Outcomes : A Pilot Feasibility Study
Brief Title: COPD Care Model on Clinical and Patient-Reported Outcomes
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 20170676-01H
Record Dates: First submitted 2017-10-10; First posted 2017-11-06 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: COPD Exacerbation
Keywords: Care Model; COPD; Exacerbations; Health Confidence Score
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthcare Professionals: Includes nurses, physicians, and allied health professionals who care for patients on the 6NW (Respirology ward) of the General campus at TOH who have implemented and worked with the COPD care pathway during the study duration.
- COPD Patients: Adult patients admitted to the 6NW (Respirology ward) of the General campus at TOH with a primary diagnosis of acute exacerbation of COPD (AECOPD). The diagnosis is based on the admitting physician's assessment of the patient in the emergency room.

SUMMARY:
This study is the first to evaluate a unique integrated care model for COPD which uses a validated clinical frailty indicator to set care goals and guide health care in hospital and in the community. The impact of this care model on patient reported outcomes, costs, and health care utilization will inform further health system re-design for patients with COPD and other chronic diseases.

DETAILED DESCRIPTION:
Background: Chronic obstructive pulmonary disease (COPD) is an incurable and progressive lung disease associated with poor quality of life, increased mortality, and high health system costs. Health system care for COPD patients is often fragmented, and patients report feeling isolated and lack the confidence in health services to address their needs.

Integrated COPD care programs attempt to address the many physical, psychosocial, and medical needs of COPD patients by bridging the gaps in care between hospital and community settings. These programs are tailored to patients with severe disease and involve self-management education sessions and sustained contact with a health care provider in the community. Evidence for the efficacy of integrated care programs is conflicting and there is limited information on which COPD patients would benefit from these programs. Prior integrated care programs have used a 'one size fits all' approach to care, where all patients receive the same interventions and treatments. There is a need for a more personalized approach to COPD care, as comorbidity burden, socioeconomic factors, and functional status also have a significant influence on health outcomes in this patient population.

Hypothesis: The investigators hypothesize that care-delivery tailored to a patient's goals and functional health status will improve patient engagement, and translate into both short and long-term improved health service outcomes.

Objectives: The objectives of this study are to: 1) Determine the feasibility of implementing a unique goal-directed COPD care model in the hospital setting, and 2) Determine the process measures and personnel required for successful replication of this care model intervention in other sites

Methods: This prospective cohort study will include 50 adult patients hospitalized for COPD exacerbation between November 2017 and May 2019. The investigators will determine the clinical frailty rating for each enrolled patient. The frailty rating will be matched with pre-specified care goals, and subsequent health care consultations and services will be arranged based upon these goals. COPD burden and 'health confidence' will be measured prior to the intervention and at 3 months following discharge, and also determine cost of hospitalization, length of stay, 30-day readmission rate, and mortality. The Wilcoxon's signed-rank test will be used to compare patient reported outcomes before and after the care intervention in the study cohort. An interrupted time series analysis will be used to determine the differences in health service outcomes between the study cohort and a random sample of hospitalized COPD patients from a contemporary period one year-prior to the care intervention.

This study will also include 26 healthcare professionals (HCPs) who work on the Respirology ward of the Ottawa Hospital, General campus during the study period. HCP's, once consented, are asked to participate in a focus group and complete a questionnaire on the COPD care Pathway.

Consent Process: Patients eligible for the study will be approached by the study respiratory nurse educator (RT), who is already part of the patients circle of care. The RT will ensure the potential participant understands the study and what it would require of them (two questionnaires: one in hospital and one during a 3-month post-discharge visit). If the patient accepts, the RT will ask them to review the Informed Consent Form and sign if they agree to participate in the study.

The clinical manager of the Respiratory ward at TOH will approach Healthcare professionals (HCPs) who work on the Respiratory ward (6NW) of TOH, General campus and have used the COPD care pathway to participate in the study. Consent forms and questionnaires will be available at the nurse's station of the Respiratory ward, of TOH General campus. The consent form requests a consent to complete a questionnaire and participate in the focus group with other HCPs. If the HCP chooses to participate, the signed informed consent is placed in one box, while the completed questionnaire is placed in another. This is to conserve anonymity of the questionnaire responses. Once focus group times and location are set, an email will be sent out by a member of the study team to inform those who consented to participate of the focus group time and location.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* COPD
* Hospitalized with a COPD exacerbations between November 2017 to May 2019 on the Respiratory ward of the Ottawa Hospital, General campus

OR

* Healthcare professional working on the Respiratory and Medicine wards of the Ottawa Hospital, General campus who used the COPD care pathway

Exclusion Criteria:

* Patients not appropriate for inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult COPD patients hospitalized with a COPD exacerbations on the Respirology or Medicine wards of the Ottawa Hospital, General campus
  and
  Healthcare professionals working on the Respiratory and Medicine wards of the Ottawa Hospital, General campus who used the COPD care pathway
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of the COPD Care Pathway on a hospital ward | 6 months from patient enrollment
  In this practical experiment, feasibility will be defined by recruitment of 50 patients (3-4 per month x 18 months) to the care pathway, with an 85% completion rate. This will be calculated using the number of completed pathway documents divided by the total number of care pathways initiated at the time of admission. Each document will be critically reviewed for completion.

SECONDARY OUTCOMES:
Qualitative Implementation Metrics - Identification of Barriers to the Care Pathway | March 2018
  Implementation of the care pathway will be evaluated by focus groups composed of health care workers (nurses, allied health professionals, and physicians) who have used the pathway. The number of focus groups planned will depend upon when data saturation is achieved. During focus groups, common themes for barriers to implementation will be identified using a-priori selected questions. Success of implementation will be considered if no significant barriers are identified through group consensus in the focus groups.
Qualitative Implementation Metrics - Healthcare Worker assessment of the Care Pathway | March 2018
  Implementation of the care pathway will also be evaluated by 2 rounds of written user survey responses from healthcare workers who used the pathway. Exit surveys have been designed to assess three domains; appropriateness of care, safety of care, and user satisfaction. Success of implementation will be considered if no significant barriers are identified through group consensus in the focus groups, and if 80% of survey responses in each domain fall into the "agree" or "strongly agree" responses.
Knowledge Translation Metrics | November 2017 to May 2019
  Knowledge translation with achievement of 80% adherence to basic COPD care guideline standards including use of appropriate antibiotics, systemic steroids, bronchodilators, venous thromboembolism prophylaxis, and advanced directives documentation. Adherence will be calculated from direct review of the order set and care pathway documents after completion.
Patient Reported 'Health Confidence' | Hospital admission to 3 months post-discharge
  Health confidence will be measured using a four-item scaled survey: 1) I know enough about my health, 2) I can look after my health, 3) I can get the right help if I need it, and 4) I am involved in decisions about me. Participants answer each of the statements with the following scale: strongly agree, agree, not sure, or disagree. Patients who report 'strongly agree' for each of the above mentioned statements are considered to have a higher level of health confidence than participants who report 'disagree'. These statements have demonstrated adequate psychometric properties and construct validity in preliminary testing (19). The health confidence survey will be administered at the start of the education session in hospital, and repeated at 3 months, during a follow-up visit.
Patient Reported 'Quality of Life' | Admission to 3 months post-discharge
  Patients quality of life can be measured with the Health Related Quality of Life Score, or 'howRu' tool which has been validated against other quality of life tools. This tool is a four-item scaled survey: 1) Pain or discomfort, 2) feeling low or worried, 3) Limited in what I can do, and 4) require help from others. Participants answer each of the statements with the following scale: none, a little, quite a lot, or extreme. Those who report 'none' for each of the above mentioned statements are considered to have a better quality of life than those who respond 'extreme'. These statements have demonstrated adequate psychometric properties and construct validity in preliminary testing (19). This survey will be administered at the start of the education session in hospital, and repeated at 3 months, during a follow-up visit.
Health Service Metrics - Length of stay in hospital | 3 months post-discharge
  Data on length of stay in hospital will be obtained from the Ottawa Hospital Data Warehouse (TOHDW). TOHDW is a relational database that captures clinical and administrative data for each unique hospital encounter.
Health Service Metrics - Cost per weighted case | 3 months post-discharge
  Data on cost per weighted case will be obtained from the Ottawa Hospital Data Warehouse (TOHDW). TOHDW is a relational database that captures clinical and administrative data for each unique hospital encounter.
Health Service Metrics - 30-day readmission | 3 months post-discharge
  Data on 30 day readmission to hospital will be obtained from the Ottawa Hospital Data Warehouse (TOHDW). TOHDW is a relational database that captures clinical and administrative data for each unique hospital encounter.
Health Service Metrics - Mortality | 6 months post-discharge
  Data on mortality in hospital will be obtained from the Ottawa Hospital Data Warehouse (TOHDW). TOHDW is a relational database that captures clinical and administrative data for each unique hospital encounter.
Health Service Metrics - Intensive Care Unit Admission | 3 months post-discharge
  Data on intensive care unit admissions will be obtained from the Ottawa Hospital Data Warehouse (TOHDW). TOHDW is a relational database that captures clinical and administrative data for each unique hospital encounter.

CONTACTS AND LOCATIONS:
Overall Officials: Sunita Mulpuru, MD, Principal Investigator — The Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital, General Campus, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2018-07-05): https://cdn.clinicaltrials.gov/large-docs/94/NCT03332394/Prot_001.pdf